CLINICAL TRIAL: NCT06450496
Title: Development of an On-line Evidence-based Positive Parenting Program for Families With Adolescents Exhibiting Mental Health Problems (Bienestar)
Brief Title: On-line Evidence-based Positive Parenting Program for Families With Adolescents Exhibiting Mental Health Problems
Acronym: Bienestar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucia Jimenez (Other)
Responsible Party: Sponsor-Investigator, Lucia Jimenez, Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2020-117363RA-I00
Record Dates: First submitted 2024-05-13; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Parenting; Wellbeing
Keywords: Effectiveness; Positive Parenting; Families; Adolescents; Mental Health; On-line Intervention; Evidence-based program; Random-control trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bienestar Program (Experimental): On-line positive parenting program
  Interventions: Behavioral: Positive parenting on-line program
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Positive parenting on-line program — Positive parenting on-line program focused on parenting and personal competences relevant for parents with adolescents exhibiting mental health problems
  Arms: Bienestar Program

SUMMARY:
This project proposes the design, implementation, and evaluation of an online psycho-educational intervention program for families of adolescents with mental health problems.

DETAILED DESCRIPTION:
Mental health problems in the child and adolescent population constitute a major challenge for society, not only because of their high prevalence but also because they undermine opportunities for the healthy development of young people, negatively impacting the wellbeing and progress of societies. Furthermore, these problems have important consequences on families of adolescents, who experience an increase in support needs, requiring effective and quality resources that allow them to adequately face the difficulties, while at the same time optimizing their parental skills to promote the development of their offspring.

Although nowadays there are more and more institutions that understand formal support to families as a social responsibility and that relies on psychoeducational programs to promote positive parenting as a beneficial strategy, the truth is that available resources aimed at covering the specific needs presented by families with adolescents with mental health problems are still scarce. Moreover, the recent emergence of the Covid-19 pandemic has resulted in even fewer evidence-based programs that are adapted to this new reality. A reality that imposes strict measures of social distance, and which generates new needs and difficulties for all families and, especially, for those who were previously in a situation of vulnerability.

In line with these approaches, and grounded in the conviction of the need to carry out applied research that is capable of transferring to society solutions derived from science and innovation, this project proposes the design, implementation, and evaluation of an online psycho-educational intervention program for families of adolescents with mental health problems.

The project presented, in line with the Spanish Law 14/2011 of 1 June on Science, Technology, and Innovation, is based on the recognition that tasks of generation, dissemination, and transference of scientific knowledge are inherent to research, as well as on the premise that the results derived from publicly funded projects should be transferred to society, contributing to the progress of citizens and meeting social challenges. In accordance with these considerations, this project aims to contribute to improving the quality of life of the families of adolescents with mental health problems by recognizing and meeting their needs, as well as optimizing parental and family skills. The achievement of this goal will involve obtaining evidence derived from empirical research that will return to society through the development and provision of an empirically validated psychoeducational intervention program aimed at promoting positive parenting in families of adolescents with mental health problems.

ELIGIBILITY:
The participants will be the caregivers (mothers or fathers) of adolescents with mental health problems of Spain. The caregiver and the target adolescent will act as respondents.

For the caregivers, the inclusion criteria are:

* Relationship with the identified patient (adolescent): Mother or father who fulfils the role of caregiver.
* They have some computer support (PC, tablet, mobile phone...) with which to carry out the program.
* Time availability to participate in the evaluation sessions.
* Motivation to participate in the program.

For the adolescents, the inclusion criteria are:

* Age between 10 and 19 years old.
* Experiencing any mental health problem.

All the inclusion criteria are requested to participate in the study.

Exclusion criteria:

Caregivers:

* Do not have an A2 Spanish language level.
* Show signs of addiction to toxic substances.

Target adolescents:

* Age less than 10 years or more than 19 years.
* Do not have an A2 Spanish language leve.

Any exclusion criteria will be considering for exclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Perceived parental role | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Me as a Parent (Hamilton et al., 2015, translation Montesdeoca, 2019)
Parental adjustment | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Global Health Questionnaire (Goldberg & Williams, 1988)

SECONDARY OUTCOMES:
Adolescent adjustment | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  The Kidscreen Questionnaire (European Kidscreen Group, 2006)
Adolescent adjustment | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Strengths and Difficulties Questionnaire (Goodman, 2001; 2022)
Satisfaction with the adolescent's life | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Satisfaction with Life Scale (Diener et al., 1985, validation Atienza et al., 2000)
Parenting styles | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Parenting Styles and Dimensions Questionnaire (Robinson et al., 2001)
Parenting styles | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Parenting Scale (Arnold et al., 1993)
Parental psychological control | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Psychological Control Scale questionnaire (Barber et al., 1996)
Parental Stress | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Parental Stress Scale (Berry & Jones; 1995, validation Oronoz et al., 2007)
Mindfulness in parenting | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  The Interpersonal Mindfulness in Parenting scale (Duncan, 2023; validation Martínez et al. 2023)
Psychological flexibility | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Acceptance and Action Questionnaire-II (Bond et al., 2011; validation Ruiz et al., 2013)
Parental psychological flexibility | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Parental Acceptance Questionnaire (Greene et al., 2015; validation Flujas-Contreras et al., 2020)
Basic Psychological Needs | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Basic Psychological Need Satisfaction and Frustration Scale (Chen et al., 2015; translation Rodríguez-Meirinhos et al., 2020)
Proactive management of basic psychological needs | At pretest, at posttest at the completion of the program (up to 2 months) and 4-to-6 months follow-up
  Need crafting questionnaire (Laporte et al., 2021; validation team, s.f.)

OTHER OUTCOMES:
Perception of usefulness of the program | At posttest atthe completion of the program (up to 2 months)
  Helpful Aspects of Therapy questionnaire adapted (Khor et al., 2021; Llewelyn et al., 1988; O'Halloran et al., 2016)
Satisfaction with the program | At posttest atthe completion of the program (up to 2 months)
  Client Satisfaction Questionnaire (Larsen et al.,1979); validation Roberts & Attkisson, 1983)
Assessment of program components | At posttest atthe completion of the program (up to 2 months)
  Parenting Online Satisfaction adapted (Suárez et al., 2018)
Usability | At posttest atthe completion of the program (up to 2 months)
  System Usability Scale (Brooke, 1996; validation Hedlefs & Villegas, 2016)
Usability | At posttest atthe completion of the program (up to 2 months)
  User Experience Questionnaire-S (Schrepp et al., 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Lucía Antolín-Suárez, PhD, Principal Investigator — University of Seville
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study not constrained by privacy or confidentiality restrictions will be stored in the publicly available repository of the University of Seville, IdUs: https://idus.us.es/.
  Further requirements by the funder of the project as well as open-access based journals will be considered.
Time Frame: Intention to publish: 31/08/2026
Access Criteria: Publicly available repository of the University of Seville, IdUs: https://idus.us.es/
URL: https://idus.us.es/